CLINICAL TRIAL: NCT06044480
Title: The Effect of Preoperative Dexamethasone on Postimplantation Syndrome After Endovascular Aneurysm Repair - Protocol for a Randomized Controlled Trial
Brief Title: Effect of Dexamethason on Postimplantation Syndrome After EVAR
Acronym: DEPOS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centro Hospitalar de Lisboa Central (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CHULC.CI.110.2020
Record Dates: First submitted 2023-06-19; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-06

CONDITIONS: Aneurysm Abdominal; Endovascular Aneurysm Repair; Postimplantation Syndrome; Dexamethasone
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dexamethasone (Active Comparator): This group of participans will be submitted to a single preoperative dose of 4 mg of dexamethasone given intravenously 30 minutes before operation.
  Interventions: Drug: Dexamethasone
- placebo (Placebo Comparator): This group of patients will be submitted to a same amount of saline solution.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Administration of a single preoperative dose of 4 mg of dexamethasone given intravenously 30 minutes before operation.
  Arms: dexamethasone
Other: Placebo — Administration of the same amount of saline solution instead of dexamethasone
  Arms: placebo

SUMMARY:
This study is a multi center double-blinded randomized controlled superiority trial, comparing the effects on postimplantatrion syndrome of a single preoperative dose of dexamethasone vs. standard treatment in endovascular aneurysm repair. Participating researchers must be vascular surgeons or vascular anesthesiologists certified by national entities. Recruitment is expected to begin in the second semester of 2023.

The trial will follow the ICH-GCP guidelines and national and international legislation and reporting will be performed according to CONSORT 2010 guidelines. Site inclusion requires hospital ethics committee approval. Written informed consent is mandatory for all patients and the information and consent forms must be approved by Institutional Ethics Committee.

DETAILED DESCRIPTION:
Post-Implantation Syndrome (PIS) consists on an inflammatory reaction after endovascular aneurysm repair of abdominal aortic aneurysms (EVAR) whose etiology and pathophysiology is still unclear, but is characterized by flu-like symptoms, with fever and elevation of analytical inflammatory parameters in the postoperative period. It is associated with a length of hospital stay and there are some studies that indicate an association with lower quality of life, increase in cardiovascular complications up to one year later and aneurysm-related complications.

PIS is defined by the presence of two criteria: tympanic temperature greater than 38ºC and CRP greater than 75 mg/L in the first three postoperative days.

Dexamethasone was the selected glucocorticoid, since it has virtually no action mineralocorticoid, has been tested in the perioperative context and is administered frequently in this context, namely at CHULC. Its use is intended to reduce symptoms associated with orotracheal extubation, pain, nausea and quality of life, without adverse effects relevant associates.

Study hypothesis: A single dose of 4mg dose of intravenous dexamethasone administered 30 minutes before surgery reduces the incidence and magnitude of PIS after EVAR.

Elegibility criteria: All the patients treated electively for a degenerative infrarenal abdominal aortic aneurysm by implantation of an endograft are eligible for this study. Patients treated for mycotic aneurysms, aortic dissections and inflammatory aneurysms are not eligible for this study, as well as patients with known inflammatory or infectious diseases and/or preoperative anti-inflammatory therapeutic.

If additional procedures, as endoanchors, proximal extension with a cuff or iliac branch device, are performed during primary EVAR, the patients should be enrolled.

Primary endpoints: The chosen primary endpoint is the occurrence of postimplantation syndrome, which is defined as fever (auricular temperature >38ºC) and elevation of CRP (> 75 mg/L), during the first 3 days after operation.

Secondary endpoints Efficacy endpoints are length of hospital stay, cardiovascular events, AAA-related complications and quality of life at 30 days and one year.

Safety endpoints relate to potential side effects of dexamethasone, as taste disturbances, hyperglycemia, flushing, rise in blood pressure, palpitations, headache, sleep isturbances,depression,euphoria, bradycardia, and cardiac decompensation in the first 30 days after operation.

ELIGIBILITY:
Inclusion Criteria:

* Elective treatment for a degenerative infrarenal abdominal aortic aneurysm by implantation of an endograft
* Additional procedures, as endoanchors, proximal extension with a cuff or iliac branch device, during primary EVAR are allowed.

Exclusion criteria:

* Mycotic aneurysms, aortic dissections and inflammatory aneurysms
* Known inflammatory or infectious diseases
* Preoperative anti-inflammatory therapeutic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Postimplantation syndrome incidence | 3 days after surgery
  Occurrence of postimplantation syndrome, which is defined as fever (auricular temperature >38ºC) and elevation of CRP (> 75 mg/L), during the first 3 days after operation.

SECONDARY OUTCOMES:
Length of hospital stay (days) | 1 year
  Efficacy outcome
cardiovascular events | 1 year
  Efficacy outcome
Rate of AAA-related complications | 1 year
  Efficacy outcome
Quality of life (EQ-5D) | 1 year
  Efficacy outcome
Safety outcomes | 30 days after surgery
  Rate of side effects of dexamethasone

IPD SHARING:
Plan to Share IPD: No